CLINICAL TRIAL: NCT05363059
Title: Army Medical University
Brief Title: Effect of Bariatric Surgery Versus Medical Therapy on Metabolic Syndrome
Acronym: EBSMTMS
Status: Recruiting | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director, Center for Hypertension and Metabolic Diseases, Department of Hypertension and Endocrinology, Daping Hospital, Third Military Medical University
Other Study IDs: EBSMTMS
Record Dates: First submitted 2022-04-18; First posted 2022-05-05 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; Medical therapy; Bariatric surgery; body mass index
MeSH Terms: conditions — Metabolic Syndrome | interventions — Hypoglycemic Agents; Antihypertensive Agents; Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BS group: The group of bariatric surgery therapy in metabolic syndrome patients.
  Interventions: Procedure: Bariatric surgery
- MT group: The group of medical therapy in metabolic syndrome patients
  Interventions: Drug: Hypoglycemic drugs

INTERVENTIONS:
Drug: Hypoglycemic drugs — drug
  Other Names: antihypertensive drugs; lipid-lowering drugs
  Groups: MT group
Procedure: Bariatric surgery — surgery
  Other Names: metabolic surgery
  Groups: BS group

SUMMARY:
Bariatric surgery (BS) is known to improve the components of metabolic syndrome (MS) in obese patients. However, few studies have evaluated the impact of bariatric surgery versus medical therapy (MT) in patients with MS, especially in patients with low body mass index (BMI). This study aimed to assess the effect of bariatric surgery on MS in patients with low BMI by comparing BS (BMI<35 kg/m2 and BMI≥35 kg/m2) with MT (BMI<35 kg/m2). A retrospective study including patients with MS undergoing bariatric surgery and medical therapy at a single institution. We follow up the 5 years effect of bariatric surgery versus medical therapy on the remission of MS, its individual components, atherosclerotic cardiovascular disease (ASCVD) risk, and medication used.

DETAILED DESCRIPTION:
1. Study design and patients

   This study aimed to compare bariatric surgery(BS) with medical therapy (MT) for the management of low BMI patients with MS, approved by the ethics committee and institutional review at our hospital. 100 patients underwent bariatric surgery and 100 patients receiving medical therapy for obesity and type 2 diabetes between 2010 and 2020 at our institution. All patients met the Chinese guidelines developed by the Chinese Society for Metabolic & Bariatric surgery (CSMBS). All patients achieve diagnostic criteria for MS, defined by the presence of at least 3 of the 5 following criteria derived from the joint interim statement (JIS) definition.
2. outcome and Data collection

   All patients follow up the change of improvement in MS and its components following bariatric surgery and medical therapy, including waist circumference, hyperglycemia, hypertension, hyperlipidemia, long-term CVD risk, and medication use
3. Treatments

3.1 BS group The bariatric surgical procedures performed included Roux-en-Y gastric bypass and sleeve gastrectomy.

3.2 MT group According to the guidelines in China, patients in the medical therapy group received glucose-lowering, lipid-lowering, and antihypertensive medications, with the following targets: glycosylated hemoglobin<7%; systolic blood pressure<140 mmHg, diastolic blood pressure<80 mmHg; low-density lipoprotein cholesterol<2.6 mmol/L; and high-density lipoprotein cholesterol>1.3 mmol/L for female or 1.0 mmol/L for male.

ELIGIBILITY:
1. Inclusion Criteria:

   * BMI<35 kg/m^2
   * Underwent bariatric surgery or medical therapy
   * Patients met the diagnostic criteria for MS, defined criteria derived from the joint interim statement (JIS)
2. Exclusion Criteria:

   * Patients who failed to follow up
   * Insulin dependent diabetes
   * congenital dementia
   * brain trauma
   * epileps
   * severe hypoglycemic coma
   * cerebrovascular disease
   * ischemic
   * heart disease
   * renal dysfunction
   * alcohol abuse
   * mental illness
   * psychoactive substance abuse
   * unwillingness to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent bariatric surgery or medical therapy for metabolic syndrome between 2010 and 2020 at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-05-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in metabolic parameters from baseline to 5 years. | baseline to 5 years
  Waist circumference(cm)
Change in metabolic parameters from baseline to 5 years. | baseline to 5 years
  body mass index(kg/m^2)

SECONDARY OUTCOMES:
Change in glycosylated hemoglobin from baseline to 5 years. | baseline to 5 years
  glycosylated hemoglobin(%)
Change in plasma glucose from baseline to 5 years. | baseline to 5 years
  Fasting plasma glucose(mmol/l),
Change in blood lipids from baseline to 5 years. | baseline to 5 years
  total cholesterol(mmol/l), triglycerides(mmol/l), high-density lipoprotein cholesterol(mmol/l), low-density lipoprotein cholesterol(mmol/l)
Changes of CVD risk | baseline to 5 years
  10-year and lifetime ASCVD risk calculated by the China-PAR equation. Evaluation metrics include sex, age, region of residence (South or North), waist circumference, total cholesterol, HDL cholesterol, systolic blood pressure, diastolic blood pressure, whether taking antihypertensive drugs, whether diabetic, whether smoker, family history of cardiovascular and cerebrovascular.
Hypoglycemic drugs use | baseline to 5 years
  The number and daily drug dose of hypoglycemic drugs
Antihypertensive drugs use | baseline to 5 years
  The number and daily drug dose of antihypertensive drugs
Lipid-lowering drugs use | baseline to 5 years
  The number and daily drug dose of lipid-lowering drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Stryker Laparoscopy, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No